CLINICAL TRIAL: NCT04628780
Title: A PHASE 1 DOSE ESCALATION AND EXPANSION STUDY TO EVALUATE SAFETY, TOLERABILITY, PHARMACOKINETIC, PHARMACODYNAMIC, AND ANTI-TUMOR ACTIVITY OF PF-07209960 IN PARTICIPANTS WITH ADVANCED OR METASTATIC SOLID TUMORS
Brief Title: Study to Test the Safety and Tolerability of PF-07209960 in Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Pfizer has made an internal business decision to not continue further development of PF-07209960. This decision was not based on safety or regulatory considerations
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C4011001; 2021-004587-10 (EudraCT Number)
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Results first posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-02

CONDITIONS: Non-small-cell Lung Cancer; Squamous Cell Carcinoma of the Head and Neck; Renal Cell Carcinoma; Urothelial Carcinoma; Colorectal Carcinoma; Ovarian Carcinoma
Keywords: PD-1; immune checkpoint inhibitor; IL-15; IL-2; cytokine; immunotherapy; Metastasis; advanced solid tumor; metastatic solid tumor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Renal Cell; Carcinoma, Transitional Cell; Colorectal Neoplasms; Ovarian Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation (Part 1) (Experimental): Participants will receive PF-07209960 at escalating dose levels
  Interventions: Biological: PF-07209960
- Dose Expansion (Part 2) - Cohort 1 (NSCLC) (Experimental): Participants with non-small cell lung cancer (NSCLC) will receive PF-07209960 at the recommended dose from Part 1
  Interventions: Biological: PF-07209960
- Dose Expansion (Part 2) - Cohort 2 (RCC) (Experimental): Participants with renal cell carcinoma (RCC) will receive PF-07209960 at the recommended dose from Part 1
  Interventions: Biological: PF-07209960
- Dose Expansion (Part 2) - Cohort 3 (UC) (Experimental): Participants with urothelial carcinoma (UC) will receive PF-07209960 at the recommended dose from Part 1
  Interventions: Biological: PF-07209960

INTERVENTIONS:
Biological: PF-07209960 — PD-1 targeted IL-15 mutein

SUMMARY:
This is a first-in-human, Phase 1, open label, multicenter, multiple dose, dose escalation and dose expansion study intended to evaluate the safety, pharmacokinetic, pharmacodynamic, and potential clinical benefit of PF-07209960, an anti-PD-1 targeting IL-15 fusion protein, in participants with selected locally advanced or metastatic solid tumors for whom no standard therapy is available, or would not be an appropriate option in the opinion of the participant and their treating physician, or participants who have refused standard therapy.

The study contains 2 parts, single agent Dose Escalation (Part 1) to determine the recommended dose of PF-07209960, followed by Dose Expansion (Part 2) in selected tumor types at the recommended dose.

ELIGIBILITY:
Inclusion Criteria:

* Histological/cytological diagnosis of selected locally advanced or metastatic solid tumor
* Demonstrated radiographic progression on most recent tumor assessment imaging
* Have ≥1 measurable lesion as defined by RECIST 1.1 that has not been previously irradiated
* Eastern Cooperative Oncology Group performance status 0-2 for Part 1 and 0-1 for Part 2
* Adequate hematologic, renal, liver, and coagulation functions
* LVEF ≥50% by echocardiogram or MUGA
* Resolved acute effects of any prior therapy
* Participants in Dose Expansion (Part 2) must have ≥2 prior lines of standard of care therapy
* Able to provide tumor tissue for submission to the Sponsor, including mandatory pre-treatment tumor biopsy (adequate archival tissue within the past 1 year is accepted in lieu of new biopsy) for all participants. Participants in Part 2 must also be able to undergo new (de novo) tumor biopsy at baseline (pre-treatment) and on-treatment biopsy until the Sponsor deems that an adequate number of biopsied samples have been received.

Exclusion Criteria:

* Known active symptomatic brain or leptomeningeal metastases requiring steroids.
* Other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ
* Major surgery or radiation therapy within 4 weeks prior to planned first dose
* Last systemic anti-cancer therapy within 4 weeks prior to planned first dose (6 weeks for mitomycin C or nitrosoureas). Participants who received anti-PD-1 therapy require an interval of 90 days prior to first dose
* Participation in other studies involving investigational drug(s) within 4 weeks prior to planned first dose
* Active and clinically significant bacterial, fungal, or viral infection; Hepatitis B or Hepatitis C infection, AIDS-related illness (HIV+ and in good immune health as defined in the protocol may be eligible)
* Active COVID-19/SARS-CoV2
* Anticoagulation with vitamin K antagonists is not allowed
* Active bleeding disorder in the past 6 months prior to first dose
* History of clinically significant severe immune mediated adverse event that was considered related to prior immune modulatory therapy and required immunosuppressive therapy (other than hormone replacement therapy)
* History of interstitial lung disease or pneumonitis
* Organ transplant requiring immunosuppressive treatment or prior allogeneic bone marrow or hematopoietic stem cell transplant
* Pregnant or breastfeeding female participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- United States (13):
  - City of Hope Investigational Drug Service (IDS), Duarte, California
  - City of Hope, Duarte, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Hematology/Oncology, Los Angeles, California
  - Santa Monica UCLA Medical Center & Orthopaedic Hospital, Santa Monica, California
  - UCLA Hematology Oncology - Santa Monica, Santa Monica, California
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - The Sarah Cannon Research Institute/Tennessee Oncology, Nashville, Tennessee
  - TriStar Centennial Medical Center, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center- Investigational Pharmacy, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Christus Santa Rosa Hospital, San Antonio, Texas
  - NEXT Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4011001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study were planned to have 2 parts: a single agent dose escalation (Part 1) followed by a dose expansion (Part 2). Due to the early termination of the study, Part 2 study was never initiated and the overall study consisted of only Part 1. The data displayed are from the Part 1 study which is the only 1 period of the study.
Pre-assignment Details: A total of 37 participants were enrolled and assigned to study treatment.
Groups:
- PF-07209960 1 mg SC: Participants with advanced or metastatic solid tumors were treated with PF-07209960 1 mg as a subcutaneous (SC) administration every 2 weeks (Q2W) for a maximum duration of 10.9 months.
- PF-07209960 3 mg SC: Participants with advanced or metastatic solid tumors were treated with PF-07209960 3 mg as a SC administration Q2W for a maximum duration of 5.1 months.
- PF-07209960 10 mg SC: Participants with advanced or metastatic solid tumors were treated with PF-07209960 10 mg as a SC administration Q2W for a maximum duration of 3.4 months.
- PF-07209960 15 mg SC: Participants with advanced or metastatic solid tumors were treated with PF-07209960 15 mg as a SC administration Q2W for a maximum duration of 5.8 months.
- PF-07209960 20 mg SC: Participants with advanced or metastatic solid tumors were treated with PF-07209960 20 mg as a SC administration Q2W for a maximum duration of 13.6 months.
- PF-07209960 30 mg SC: Participants with advanced or metastatic solid tumors were treated with PF-07209960 30 mg as a SC administration Q2W for a maximum duration of 12.6 months.
Period: Overall Study
Arm/Group | PF-07209960 1 mg SC | PF-07209960 3 mg SC | PF-07209960 10 mg SC | PF-07209960 15 mg SC | PF-07209960 20 mg SC | PF-07209960 30 mg SC
Started | 4 | 4 | 4 | 3 | 16 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 4 | 4 | 3 | 16 | 6
Not completed — Death | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 2 | 0
Not completed — Progressive disease | 2 | 2 | 2 | 3 | 9 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 0 | 3 | 1
Not completed — Global deterioration of health status | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-07209960 1 mg SC | PF-07209960 3 mg SC | PF-07209960 10 mg SC | PF-07209960 15 mg SC | PF-07209960 20 mg SC | PF-07209960 30 mg SC | Total
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 16 | 6 | 37
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Mean | 67.0 (14.49) | 60.5 (15.33) | 60.8 (7.41) | 54.0 (4.58) | 56.6 (11.14) | 54.8 (13.92) | 58.1 (11.65)
Age, Customized [Count of Participants; unit: Participants]
  18-44 years | 0 | 0 | 0 | 0 | 3 | 1 | 4
  45-64 years | 2 | 3 | 3 | 3 | 10 | 3 | 24
  >=65 years | 2 | 1 | 1 | 0 | 3 | 2 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 1 | 9 | 1 | 17
  Male | 2 | 2 | 2 | 2 | 7 | 5 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 0 | 5 | 1 | 9
  Not Hispanic or Latino | 2 | 3 | 4 | 3 | 11 | 4 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 3 | 4 | 3 | 12 | 5 | 30
  Asian | 0 | 0 | 0 | 0 | 3 | 0 | 3
  Not reported | 1 | 1 | 0 | 0 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: For the purpose of dose escalation, any of the following adverse events were classified as DLTs: Occur in the first cycle of treatment, or within 28 days after the start of the study treatment; and were at least possibly related to PF-07209960; A participant was classified as DLT evaluable if he/she experienced a DLT or if he/she otherwise in the absence of a DLT received 2 doses of the study intervention during Cycle 1 and had received all scheduled safety assessments during the DLT window. If a participant failed to meet these criteria, he/she might be replaced. Monitoring for DLTs occurred during Part 1.
Time Frame: Cycle 1 (28 days)
Population: The DLT analysis set was a subset of the safety analysis set. A participant was classified as DLT-evaluable if he/she experienced a DLT or received 100% of the planned doses and had received all scheduled safety assessments during the DLT window.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07209960 1 mg SC | PF-07209960 3 mg SC | PF-07209960 10 mg SC | PF-07209960 15 mg SC | PF-07209960 20 mg SC | PF-07209960 30 mg SC
Number analyzed (Participants) | 4 | 3 | 4 | 2 | 10 | 4
Participants | 0 | 0 | 0 | 0 | 3 | 3

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Adverse event (AE) was any untoward medical occurrence in a participant who received any study drug without regard to possibility of causal relationship. TEAEs were those events with onset dates occurring during the on-treatment period. On-treatment period was defined as time from first dose of any study treatment and up to 90 days after last dose or start day of new anti-cancer drug therapy minus 1 day, whichever occurred first. Treatment-related AEs were those related to any study drug (ie, at least one of the study drugs).
Time Frame: From start of the treatment until a minimum of 90 days after the last dose of study intervention (maximum up to 16.6 months)
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07209960 1 mg SC | PF-07209960 3 mg SC | PF-07209960 10 mg SC | PF-07209960 15 mg SC | PF-07209960 20 mg SC | PF-07209960 30 mg SC
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 16 | 6
Participants
  Participants with all-causality TEAEs | 4 | 4 | 3 | 3 | 16 | 6
  Participants with treatment-related TEAEs | 1 | 2 | 2 | 3 | 14 | 6

3. Primary Outcome: Number of Participants With Maximum Grade 3 or 4 TEAEs
Description: AE was any untoward medical occurrence in a participant who received any study drug without regard to possibility of causal relationship. TEAEs were those events with onset dates occurring during the on-treatment period. On-treatment period was defined as time from first dose of any study treatment and up to 90 days after last dose or start day of new anti-cancer drug therapy minus 1 day, whichever occurred first. TEAEs were graded by the investigator using National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) version 5.0 as Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = death. In this outcome measure, number of participants with Maximum Grade 3 or 4 TEAEs were reported.
Time Frame: as for outcome 2
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07209960 1 mg SC | PF-07209960 3 mg SC | PF-07209960 10 mg SC | PF-07209960 15 mg SC | PF-07209960 20 mg SC | PF-07209960 30 mg SC
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 16 | 6
Participants
  Participants with Maximum Grade 3 or 4 TEAEs (all-causality) | 3 | 2 | 1 | 1 | 11 | 5
  Participants with Maximum Grade 3 or 4 TEAEs (treatment-related) | 0 | 0 | 1 | 2 | 8 | 5

4. Primary Outcome: Number of Participants With TEAEs Leading to Death
Description: TEAEs were those events with onset dates occurring during the on-treatment period.
Time Frame: as for outcome 2
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07209960 1 mg SC | PF-07209960 3 mg SC | PF-07209960 10 mg SC | PF-07209960 15 mg SC | PF-07209960 20 mg SC | PF-07209960 30 mg SC
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 16 | 6
Participants
  Participants with all-causality TEAEs leading to death | 1 | 1 | 0 | 1 | 2 | 1
  Participants with treatment-related TEAEs leading to death | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Serious TEAEs
Description: TEAEs were those events with onset dates occurring during the on-treatment period. On-treatment period was defined as time from first dose of any study treatment until a minimum of 90 days after the last dose of study intervention. Treatment-related AEs were those related to any study drug (ie, at least one of the study drugs). A serious TEAE was any untoward medical occurrence that at any dose resulted in any of following outcomes/considered to be an important medical event: death; life-threatening experience (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); congenital anomaly/birth defect.
Time Frame: as for outcome 2
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07209960 1 mg SC | PF-07209960 3 mg SC | PF-07209960 10 mg SC | PF-07209960 15 mg SC | PF-07209960 20 mg SC | PF-07209960 30 mg SC
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 16 | 6
Participants
  Participants with all-causality serious TEAEs | 3 | 3 | 1 | 1 | 13 | 5
  Participants with treatment-related serious TEAEs | 0 | 1 | 0 | 1 | 7 | 4

6. Primary Outcome: Number of Participants Discontinued From Study Due to TEAEs
Description: Participants who had an AE record that indicated that the AE caused the participant to be discontinued from the study. TEAEs were those events with onset dates occurring during the on-treatment period. On-treatment period was defined as time from first dose of any study treatment until a minimum of 90 days after the last dose of study intervention. Treatment-related AEs were those related to any study drug (ie, at least one of the study drugs).
Time Frame: as for outcome 2
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07209960 1 mg SC | PF-07209960 3 mg SC | PF-07209960 10 mg SC | PF-07209960 15 mg SC | PF-07209960 20 mg SC | PF-07209960 30 mg SC
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 16 | 6
Participants
  Participants discontinued from study due to all-causality TEAEs | 0 | 1 | 0 | 1 | 2 | 1
  Participants discontinued from study due to treatment-related TEAEs | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With New or Worsening Hematology Laboratory Test Results to Grade >=1 During the On-Treatment Period
Description: The number of participants with newly occurring or worsening hematology abnormalities during the on-treatment period were summarized by worst grade on-treatment. NCI-CTCAE criteria version 5.0 is used. As per NCI CTCAE toxicity grading v5.0, Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = death.
Time Frame: as for outcome 2
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07209960 1 mg SC | PF-07209960 3 mg SC | PF-07209960 10 mg SC | PF-07209960 15 mg SC | PF-07209960 20 mg SC | PF-07209960 30 mg SC
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 16 | 6
Participants
  Activated partial thromboplastin time prolonged | 0 | 1 | 1 | 2 | 13 | 5
  Anemia | 3 | 4 | 4 | 3 | 15 | 6
  Fibrinogen decreased | 0 | 0 | 0 | 0 | 4 | 2
  Hemoglobin increased | 0 | 0 | 0 | 0 | 0 | 0
  INR increased | 0 | 1 | 1 | 1 | 8 | 4
  Leukocytosis | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased | 3 | 3 | 4 | 3 | 16 | 6
  Lymphocyte count increased | 1 | 0 | 1 | 1 | 3 | 1
  Neutrophil count decreased | 0 | 0 | 1 | 1 | 3 | 3
  Platelet count decreased | 1 | 2 | 2 | 2 | 10 | 5
  White blood cell decreased | 1 | 0 | 1 | 3 | 6 | 4

8. Primary Outcome: Number of Participants With New or Worsening Hematology Laboratory Test Results to Grade >=3 During the On-Treatment Period
Description: as for outcome 7
Time Frame: as for outcome 2
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07209960 1 mg SC | PF-07209960 3 mg SC | PF-07209960 10 mg SC | PF-07209960 15 mg SC | PF-07209960 20 mg SC | PF-07209960 30 mg SC
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 16 | 6
Participants
  Activated partial thromboplastin time prolonged | 0 | 0 | 0 | 0 | 0 | 0
  Anemia | 0 | 0 | 1 | 1 | 4 | 1
  Fibrinogen decreased | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased | 0 | 0 | 0 | 0 | 0 | 0
  INR increased | 0 | 0 | 0 | 0 | 2 | 1
  Leukocytosis | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased | 0 | 2 | 2 | 3 | 16 | 6
  Lymphocyte count increased | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil count decreased | 0 | 0 | 0 | 0 | 1 | 1
  Platelet count decreased | 0 | 0 | 0 | 0 | 0 | 1
  White blood cell decreased | 0 | 0 | 0 | 0 | 0 | 1

9. Primary Outcome: Number of Participants With New or Worsening Chemistry Laboratory Test Results to Grade >=1 During the On-Treatment Period
Description: The number of participants with newly occurring or worsening chemistry abnormalities during the on-treatment period were summarized by worst grade on-treatment. NCI-CTCAE criteria version 5.0 is used. As per NCI CTCAE toxicity grading v5.0, Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = death.
Time Frame: as for outcome 2
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07209960 1 mg SC | PF-07209960 3 mg SC | PF-07209960 10 mg SC | PF-07209960 15 mg SC | PF-07209960 20 mg SC | PF-07209960 30 mg SC
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 16 | 6
Participants
  Alanine aminotransferase increased | 0 | 1 | 2 | 0 | 8 | 5
  Alkaline phosphatase increased | 1 | 1 | 2 | 3 | 8 | 4
  Aspartate aminotransferase increased | 2 | 1 | 3 | 3 | 9 | 4
  Blood bilirubin increased | 0 | 0 | 0 | 1 | 8 | 2
  Creatinine increased | 3 | 0 | 2 | 2 | 8 | 4
  Hypercalcemia | 3 | 0 | 0 | 1 | 3 | 2
  Hyperkalemia | 2 | 0 | 0 | 1 | 1 | 1
  Hypermagnesemia | 1 | 0 | 0 | 0 | 0 | 0
  Hypernatremia | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia | 3 | 1 | 2 | 3 | 14 | 5
  Hypocalcemia | 0 | 0 | 0 | 0 | 2 | 0
  Hypoglycemia | 1 | 1 | 0 | 0 | 3 | 1
  Hypokalemia | 1 | 0 | 1 | 1 | 12 | 1
  Hypomagnesemia | 3 | 0 | 1 | 3 | 4 | 4
  Hyponatremia | 2 | 2 | 2 | 3 | 15 | 5

10. Primary Outcome: Number of Participants With New or Worsening Chemistry Laboratory Test Results to Grade >=3 During the On-Treatment Period
Description: as for outcome 9
Time Frame: as for outcome 2
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07209960 1 mg SC | PF-07209960 3 mg SC | PF-07209960 10 mg SC | PF-07209960 15 mg SC | PF-07209960 20 mg SC | PF-07209960 30 mg SC
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 16 | 6
Participants
  Alanine aminotransferase increased | 0 | 0 | 0 | 0 | 1 | 0
  Alkaline phosphatase increased | 0 | 0 | 1 | 0 | 0 | 0
  Aspartate aminotransferase increased | 0 | 0 | 0 | 0 | 2 | 0
  Blood bilirubin increased | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine increased | 0 | 0 | 0 | 1 | 1 | 0
  Hypercalcemia | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia | 0 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia | 0 | 0 | 0 | 0 | 0 | 1
  Hypocalcemia | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia | 0 | 0 | 0 | 0 | 1 | 0
  Hypokalemia | 1 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia | 0 | 0 | 0 | 2 | 1 | 2

11. Secondary Outcome: Percentage of Participants With Objective Response (OR) as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: Objective Response Rate (ORR) is defined as the percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR) per RECIST version 1.1. CR: Complete disappearance of all target and non-target lesions with the exception of nodal disease; all target and non-target nodes must decrease to normal size (short axis <10 mm); all lesions must be assessed. PR: Greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions; all target lesions must be assessed. Non-target PR lesions must be non-progressive disease (PD), where PD is unequivocal progression of pre-existing lesions.
Time Frame: From start of the treatment until disease progression or discontinuation from study or death due to any cause, whichever occurred first (maximum up to 14.5 months)
Population: Response evaluable set included all participants who received at least one dose of study treatment and had measurable disease at baseline and at least one post baseline disease assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PF-07209960 1 mg SC | PF-07209960 3 mg SC | PF-07209960 10 mg SC | PF-07209960 15 mg SC | PF-07209960 20 mg SC | PF-07209960 30 mg SC
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 11 | 5
Percentage of participants | 0 [0.0 to 70.8] | 0 [0.0 to 60.2] | 0 [0.0 to 70.8] | 0 [0.0 to 70.8] | 9.1 [0.2 to 41.3] | 20.0 [0.5 to 71.6]

12. Secondary Outcome: Number of Participants by Antidrug Antibody (ADA) Categories
Description: Immunogenicity blood samples were assayed for ADA using a validated assay. The sample analysis followed a tiered approach of screening, confirmation, and titer determination. Samples tested positive for ADA were further analyzed for neutralizing antibodies (Nab) using a validated assay. Baseline is defined as pre-dose measurement on Day 1. n=Number of ADA evaluable participants with positive ADA at baseline; n1=Number of ADA evaluable participants with positive ADA at baseline but did not become boosted post-treatment; n2=Number of ADA-positive participants (treatment-induced or treatment-boosted).
Time Frame: on Day 1,15 and 22 of Cycle 1, on Day 1 of Cycles 2-9, and then on Day 1 of Cycles 12, 15, and at the end of treatment (EOT)
Population: Immunogenicity analysis set includes all enrolled participants who receive at least one dose of study treatment and have at least one sample tested for ADA. Number of participants analyzed = Number of participants with >=1 post-treatment ADA result (N1).
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07209960 1 mg SC | PF-07209960 3 mg SC | PF-07209960 10 mg SC | PF-07209960 15 mg SC | PF-07209960 20 mg SC | PF-07209960 30 mg SC
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 14 | 5
Participants
  Evaluable participants with pre-existing antibody, n/N1 | 1 | 0 | 4 | 0 | 6 | 1
  Baseline-positive participants with non-boosted antibody response, n1/N1 | 0 | 0 | 1 | 0 | 1 | 0
  Overall Incidence, n2/N1 | 4 | 3 | 3 | 3 | 13 | 5
  Treatment-induced | 3 | 3 | 0 | 3 | 8 | 4
  Treatment-boosted | 1 | 0 | 3 | 0 | 5 | 1

13. Secondary Outcome: Number of Participants by ADA Against Endogenous IL-15 Wild-type Categories
Description: Immunogenicity blood samples were assayed for ADA using a validated assay. The sample analysis followed a tiered approach of screening, confirmation, and titer determination. Samples tested positive for ADA were further analyzed for neutralizing antibodies (Nab) using a validated assay. Baseline is defined as pre-dose measurement on Day 1. n=Number of ADA evaluable participants with positive ADA at baseline; n2=Number of ADA-positive participants.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07209960 1 mg SC | PF-07209960 3 mg SC | PF-07209960 10 mg SC | PF-07209960 15 mg SC | PF-07209960 20 mg SC | PF-07209960 30 mg SC
Number analyzed (Participants) | 4 | 2 | 3 | 3 | 13 | 5
Participants
  Evaluable participants with pre-existing antibody, n/N1 | 1 | 0 | 0 | 0 | 0 | 0
  Overall Incidence, n2/N1 | 1 | 1 | 1 | 1 | 4 | 1

14. Secondary Outcome: Number of Participants by Anti-IL-15 Wild Type NAb Categories
Description: Immunogenicity blood samples were assayed for ADA using a validated assay. The sample analysis followed a tiered approach of screening, confirmation, and titer determination. Samples tested positive for ADA were further analyzed for neutralizing antibodies (NAb) using a validated assay. Baseline is defined as pre-dose measurement on Day 1. N1=Number of participants with ≥ 1 post-treatment NAb result; n=Number of NAb evaluable participants with positive NAb at baseline; n2=Number of NAb-positive participants (treatment induced).
Time Frame: as for outcome 12
Population: Immunogenicity analysis set includes all enrolled participants who receive at least one dose of study treatment and have at least one sample tested for ADA. Number of participants analyzed = Number of participants with >=1 post-treatment NAb result (N1).
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07209960 1 mg SC | PF-07209960 3 mg SC | PF-07209960 10 mg SC | PF-07209960 15 mg SC | PF-07209960 20 mg SC | PF-07209960 30 mg SC
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 14 | 5
Participants
  Evaluable participants with pre-existing antibody, n/N1 | 0 | 0 | 0 | 0 | 0 | 0
  Overall Incidence, n2/N1 | 1 | 2 | 1 | 1 | 1 | 2

15. Secondary Outcome: Time to Progression (TTP) in Participants With Progressive Disease Based on Investigator Assessment
Description: TTP is defined as the time from start date of treatment to the date of the first documentation of PD or censoring. TTP is similar to PFS except that death is not treated as an event and is censored. Both new anti-cancer therapy given prior to PD and no PD by the end of follow-up are censoring events
Time Frame: Baseline through up to 2 years or until disease progression
Population: The full analysis set included all enrolled participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PF-07209960 1 mg SC | PF-07209960 3 mg SC | PF-07209960 10 mg SC | PF-07209960 15 mg SC | PF-07209960 20 mg SC | PF-07209960 30 mg SC
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 16 | 6
Months | 3.7 [1.4 to NA] — Upper limit of 95% CI was not reached due to fewer number of participants with event. | 2.8 [2.7 to NA] — Upper limit of 95% CI was not reached due to fewer number of participants with event. | 3.8 [1.9 to NA] — Upper limit of 95% CI was not reached due to fewer number of participants with event. | 1.6 [1.5 to NA] — Upper limit of 95% CI was not reached due to fewer number of participants with event. | 1.8 [1.6 to 3.7] | 2.0 [0.9 to NA] — Upper limit of 95% CI was not reached due to fewer number of participants with event.

16. Secondary Outcome: Duration of Response (DOR) Based on Investigator Assessment in Participants With Confirmed Response
Description: DOR is defined as the time from first documentation of CR or PR to date of first documentation of objective progression, or death due to any cause, or time of censoring, whichever occurred first.
Time Frame: Baseline through up to 2 years or until disease progression
Population: The full analysis set included all enrolled participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PF-07209960 20 mg SC | PF-07209960 30 mg SC
Number analyzed (Participants) | 1 | 1
Months | 9.5 [NA to NA] — Only 1 participant had DOR record | 3 [NA to NA] — Only 1 participant had DOR record

17. Secondary Outcome: Progression-Free Survival (PFS) Based on Investigator Assessment in Participants
Description: PFS is defined as time from start date of treatment to the date of first documentation of PD or death due to any cause, or censoring, whichever occurred first. Both new anti-cancer therapy given prior to PD or death and no PD by the end of follow-up are censoring events.
Time Frame: Baseline through up to 2 years or until disease progression
Population: The full analysis set includes all enrolled participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PF-07209960 1 mg SC | PF-07209960 3 mg SC | PF-07209960 10 mg SC | PF-07209960 15 mg SC | PF-07209960 20 mg SC | PF-07209960 30 mg SC
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 16 | 6
Months | 2.8 [1.4 to NA] — Upper limit of 95% CI was not reached due to fewer number of participants with event. | 2.8 [2.7 to NA] — Upper limit of 95% CI was not reached due to fewer number of participants with event. | 3.8 [1.9 to NA] — Upper limit of 95% CI was not reached due to fewer number of participants with event. | 1.6 [1.5 to NA] — Upper limit of 95% CI was not reached due to fewer number of participants with event. | 1.8 [1.4 to 3.5] | 2.0 [0.9 to NA] — Upper limit of 95% CI was not reached due to fewer number of participants with event.

18. Secondary Outcome: Percentage of Participants With Disease Control Based on Investigator Assessment
Description: Disease control rate (DCR) is defined as the percentage of participants with a BOR of CR, PR, non-CR/non-PD or SD.
Time Frame: From start of the treatment until disease progression or death due to any cause, whichever occurred first (maximum up to 2 years approximately)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | PF-07209960 1 mg SC | PF-07209960 3 mg SC | PF-07209960 10 mg SC | PF-07209960 15 mg SC | PF-07209960 20 mg SC | PF-07209960 30 mg SC
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 11 | 5
Percentage of Participants | 66.7 [9.4 to 99.2] | 75.0 [19.4 to 99.4] | 66.7 [9.4 to 99.2] | 0 [0.0 to 70.8] | 45.5 [16.7 to 76.6] | 40.0 [5.3 to 85.3]

ADVERSE EVENTS:
Time Frame: AEs are reported based on the on-treatment period (from first dose to 90 days post-last dose or start of new anti-cancer therapy - 1 day) for a maximum duration of 16.6 months.
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. Safety set was evaluated. The safety analysis set included all participants who received at least 1 dose of study drug. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | PF-07209960 1 mg SC | PF-07209960 3 mg SC | PF-07209960 10 mg SC | PF-07209960 15 mg SC | PF-07209960 20 mg SC | PF-07209960 30 mg SC
All-Cause Mortality (participants affected / at risk) | 1/4 | 1/4 | 1/4 | 1/3 | 3/16 | 1/6
Serious Adverse Events (participants affected / at risk) | 3/4 | 3/4 | 1/4 | 1/3 | 13/16 | 5/6
Other Adverse Events (participants affected / at risk) | 4/4 | 2/4 | 3/4 | 3/3 | 16/16 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-07209960 1 mg SC (N=4) | PF-07209960 3 mg SC (N=4) | PF-07209960 10 mg SC (N=4) | PF-07209960 15 mg SC (N=3) | PF-07209960 20 mg SC (N=16) | PF-07209960 30 mg SC (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Disease progression (General disorders) | 1 | 0 | 0 | 1 | 1 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 3 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 7 | 4
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 1
Bladder perforation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-07209960 1 mg SC (N=4) | PF-07209960 3 mg SC (N=4) | PF-07209960 10 mg SC (N=4) | PF-07209960 15 mg SC (N=3) | PF-07209960 20 mg SC (N=16) | PF-07209960 30 mg SC (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 4 | 2
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 2 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 3 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Lip disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 7 | 2
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 1 | 1 | 3 | 1
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 2 | 1 | 6 | 3
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Injection site reaction (General disorders) | 1 | 0 | 0 | 3 | 5 | 2
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 2 | 1 | 1
Pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 8 | 2
Swelling face (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 1 | 2 | 5 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Herpes simplex reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Lymph gland infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pyuria (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Stoma site reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 3 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 3 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2
Interleukin level increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 3 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 2
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 3 | 3
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 2
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 4 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 3
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 2
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 3 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Penile swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 6 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2 | 4 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 0
Pharyngeal paraesthesia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 5 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 1
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was planned to have 2 parts: a single agent dose escalation (Part 1) followed by a dose expansion (Part 2).

Due to the early termination of the study, Part 2 study was never initiated and the overall study consisted of only Part 1. The data displayed are from the Part 1 study which is the only 1 period of the study. Besides, the pharmacokinetic (PK) endpoints of this study were not conducted. Therefore no results of PK parameters are displayed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/80/NCT04628780/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT04628780/SAP_001.pdf